CLINICAL TRIAL: NCT03485742
Title: Statin Eligibility Prior to Myocardial InfarCtion in Jordanians
Brief Title: Statin Eligibility Prior to Myocardial InfarCtion
Acronym: StatinEPIC
Status: Terminated | Type: Observational
Why Stopped: We recruited a target number (740 patients) earlier than the expected day of copletion
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: JCCStatinEpic2018
Record Dates: First submitted 2018-03-17; First posted 2018-04-02 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Statins; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention. Collection of data on statin eligibility in patients admitted with MI

SUMMARY:
The study (Statin Eligibility Prior to myocardial infarction (MI) in Jordanians, StatinEPIC) is

1. Cross sectional
2. Non interventional
3. One encounter per patient. No follow up. It addresses a major issue of primary prevention in Jordanians especially the young population, namely the issue of lipid lowering agents before sustaining an acute MI. A recent study in USA showed that 50% of patients who sustained MI were not eligible to statins had they been evaluated before the heart attack. It is largely unknown if a larger percentage of Middle Eastern patients who sustain a heart attack would be eligible to receive lipid lowering agents.
4. The PI will overlook the whole process. Dr Ahmad Tamari, the assistant to the PI will asses this whole process of data collection, management and manuscript drafting.

DETAILED DESCRIPTION:
Statins, when use as primary cardiovascular prevention strategy, have been shown to lower future acute cardiovascular events, especially myocardial infarction. However the use of statins in this context (i.e., primary prevention) is governed by guidelines that limit the use of statins to four high risk populations: (1) hose with known cardiovascular disease, (2) those with low-density lipoprotein cholesterol (LDL-C) levels 190 mg/dl or above, (3) diabetics with LDL-C levels 70-189 mg/dl, and (4) those with an estimated 10-year atherosclerotic cardiovascular disease risk score of 7.5% or more.

Unfortunately, some individuals are still at risk of sustaining MI despite the fact that they do not fit into one of these four high risk groups eligible for statins.

StainEPIC will enroll consecutive patients admitted with MI who are not on statins to examine their eligibility for these medications based on the AHA/ACC guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted with MI, age 30 to 75
* known lipid profile

Exclusion Criteria:

* on statin before enrollment

Ages: 30 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, female
Study Population: Patients aged 30 to 75 years admitted with MI (ST elevation and non ST elevation) who are not receiving statins prior to admission will be evaluated for potential eligibility had they been evaluated prior to admission with MI.
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Eligible patients for statin therapy | Within 24 hour of enrollment
  The primary outcome is to calculate the percentage of enrolled patients who do meet the AHA/ACC Guidelines for receiving statins as a primary prevention measure.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine Obeidat, MS, Study Director — Hashemmeyyeh University School of Medicine, Zarka, Jordan; Ayman J Hammoudeh, MD, FACC, Principal Investigator — Istishari Hospital, Department of Cardiology, Amman, Jordan
Locations (5):
- Jordan (5):
  - Istishari Hospital, Amman
  - The University of Jordan, Amman
  - Jordan Hospital, Amman
  - Khalidi Hospital & Medical Center, Amman
  - King Abdullah University Hospital, Irbid

IPD SHARING:
Plan to Share IPD: No
All IPD files will be available for all study researchers: clinical data, lipid profile data, 10 year risk score data, statin eligibility data.